CLINICAL TRIAL: NCT06241508
Title: The Modulatory Effect of Low-intensity Priming Intermittent Theta Burst Stimulation on Motor Cortex Poststroke: a Concurrent TMS-EEG Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20231104003
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: stroke; transcranial magnetic stimulation; theta burst stimulation; neuroplasticity; motor learning
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-intensity priming intermittent theta burst stimulation (Experimental): Theta burst stimulation (TBS) is a potent form of repetitive transcranial magnetic stimulation (rTMS). Standard 600-pulse intermittent theta burst stimulation (iTBS) can enhance the corticomotor excitability, whereas standard 600-pulse continuous theta burst stimulation (cTBS) can suppress the corticomotor excitability. Sham stimulation uses an extreme low stimulation intensity which will not influence with corticomotor excitability.
  In the present study, real stimulation will be delivered in an intensity of 55% (low-intensity) or 70% (conventional intensity) individual resting motor threshold while sham stimulation will be delivered in an intensity of 20% (ineffective) individual resting motor threshold.
  Low-intensity priming intermittent theta burst stimulation will use a session of 55% RMT cTBS followed by a session of 70% RMT iTBS. Both sessions will be applied to the ipsilesional primary motor cortex.
  Interventions: Device: Transcranial magnetic stimulation
- Conventional intensity priming intermittent theta burst stimulation (Experimental): Theta burst stimulation (TBS) is a potent form of repetitive transcranial magnetic stimulation (rTMS). Standard 600-pulse intermittent theta burst stimulation (iTBS) can enhance the corticomotor excitability, whereas standard 600-pulse continuous theta burst stimulation (cTBS) can suppress the corticomotor excitability. Sham stimulation uses an extreme low stimulation intensity which will not influence with corticomotor excitability.
  In the present study, real stimulation will be delivered in an intensity of 55% (low-intensity) or 70% (conventional intensity) individual resting motor threshold while sham stimulation will be delivered in an intensity of 20% (ineffective) individual resting motor threshold.
  Conventional intensity priming intermittent theta burst stimulation will use a session of 70% RMT cTBS followed by a session of 70% RMT iTBS. Both sessions will be applied to the ipsilesional primary motor cortex.
  Interventions: Device: Transcranial magnetic stimulation
- Standard, nonpriming intermittent theta burst stimulation (Active Comparator): Theta burst stimulation (TBS) is a potent form of repetitive transcranial magnetic stimulation (rTMS). Standard 600-pulse intermittent theta burst stimulation (iTBS) can enhance the corticomotor excitability, whereas standard 600-pulse continuous theta burst stimulation (cTBS) can suppress the corticomotor excitability. Sham stimulation uses an extreme low stimulation intensity which will not influence with corticomotor excitability.
  In the present study, real stimulation will be delivered in an intensity of 55% (low-intensity) or 70% (conventional intensity) individual resting motor threshold while sham stimulation will be delivered in an intensity of 20% (ineffective) individual resting motor threshold.
  Nonpriming priming intermittent theta burst stimulation will use a session of 20% RMT cTBS followed by a session of 70% RMT iTBS. Both sessions will be applied to the ipsilesional primary motor cortex.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — A standard 600-pulse TBS [16] will be administrated using a MagPro X100 stimulator (MagVenture, Denmark) and a 65-mm figure-of-eight coil. The measurement of the motor hotspot and individual RMT will be in accordance with our established methodology [3, 9]. For patients with stroke, the intensity of real stimulation will be 55% or 70% RMT of the unaffected M1 [17], depending on their assigned condition. Sham stimulation will be delivered using the same coil with 20% RMT of the unaffected M1 [4, 6]. The priming and conditioning sessions will be delivered to the ipsilesional M1 sequentially. In line with previous works, the interval between them will be 10 minutes [2, 3]. For healthy adults, the stimulation will be applied exclusively to the non-dominant (right) M1.

SUMMARY:
Background: The optimization of the intensity of priming theta burst stimulation increases the probability of success in a randomized controlled trial. We hypothesize that priming intermittent theta burst stimulation (iTBS) with a low-intensity continuous theta burst stimulation (cTBS) will yield superior effects than our original priming protocol in healthy adults and patients after stroke.

Methods: 20 stroke patients will undergo three separate experimental conditions: a low-intensity priming stimulation (55% resting motor threshold [RMT] cTBS+70% RMT iTBS), a conventional-intensity priming stimulation (70% RMT cTBS+70% RMT iTBS), and a nonpriming control. The alterations in cortical excitation/inhibition and its impacts on motor behaviors will be evaluated following stimulation.

Significance: The findings will inform future clinical trials investigating the optimized priming iTBS in promoting poststroke recovery.

DETAILED DESCRIPTION:
Background: The optimization of the intensity of priming theta burst stimulation increases the probability of success in a randomized controlled trial. We hypothesize that priming intermittent theta burst stimulation (iTBS) with a low-intensity continuous theta burst stimulation (cTBS) will yield superior effects than our original priming protocol in healthy adults and patients after stroke.

Methods: 20 stroke patients will undergo three separate experimental conditions: a low-intensity priming stimulation (55% resting motor threshold [RMT] cTBS+70% RMT iTBS), a conventional-intensity priming stimulation (70% RMT cTBS+70% RMT iTBS), and a nonpriming control. The alterations in cortical excitation/inhibition and its impacts on motor behaviors will be evaluated following stimulation.

Significance: The findings will inform future clinical trials investigating the optimized priming iTBS in promoting poststroke recovery.

ELIGIBILITY:
Inclusion Criteria:

* (1) have a diagnosis of ischemic or hemorrhagic stroke, with time after stroke onset≥6 months;
* (2) aged between 18 and 80 years old;
* (3) with residual upper limb functions from 2-7 levels in the Functional Test for the Hemiplegic Upper Extremity, i.e., moderately impaired overall upper extremity functions.
* (4) able to give informed written consent to participate in the study.

Exclusion Criteria:

* (1) any contraindications to TMS (screened by the safety checklist by Rossi [12]); -
* (2) any concomitant neurological disease;
* (3) any sign of moderate-to-severe cognitive problems, i.e., Montreal cognitive assessment (MoCA)<19/30
* (4) Modified Ashworth score>2 in hand, wrist or elbow extensor muscle in the hemiparetic upper extremity.

In addition, a group of age-matched, right-hand dominant healthy adults without any known neurological diseases will be enrolled. Healthy adults with any contraindications to TMS will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
The isometric force control task | Baseline
  Force data will be collected using a load cell (Force sensor ZNHM, Chino sensor, China). To assess maximal voluntary contraction (MVC) of the hand grip, three trials will be conducted using both paretic and nonparetic hands (or the dominant and non-dominant hands for healthy controls). Subsequently, separate tests will be performed to measure submaximal isometric force at 20% and 50% of the maximal voluntary force (MVF). Each trial will last for 20 seconds, with a 60-second intertrial interval to prevent fatigue. A total of 5 trials will be conducted for each level of muscle contraction. Muscle strength will be evaluated by calculating the mean force output, while the variability of force control will be assessed by calculating the coefficient of variation of force, i.e., the standard deviation of force/mean force output × 100%.
The isometric force control task | 15-min after completion of stimulation sessions
  Force data will be collected using a load cell (Force sensor ZNHM, Chino sensor, China). To assess maximal voluntary contraction (MVC) of the hand grip, three trials will be conducted using both paretic and nonparetic hands (or the dominant and non-dominant hands for healthy controls). Subsequently, separate tests will be performed to measure submaximal isometric force at 20% and 50% of the maximal voluntary force (MVF). Each trial will last for 20 seconds, with a 60-second intertrial interval to prevent fatigue. A total of 5 trials will be conducted for each level of muscle contraction. Muscle strength will be evaluated by calculating the mean force output, while the variability of force control will be assessed by calculating the coefficient of variation of force, i.e., the standard deviation of force/mean force output × 100%.
Transcranial magnetic stimulation-evoked potential | Baseline
  Single pulses evoked an initial response in electroencephalogram, followed by a series of time- and phase-locked positive and negative deflections which could spread to the connected brain areas. The evoked potential is called transcranial magnetic stimulation-evoked potential.
Transcranial magnetic stimulation-evoked potential | 5-min after completion of stimulation sessions
  Single pulses evoked an initial response in electroencephalogram, followed by a series of time- and phase-locked positive and negative deflections which could spread to the connected brain areas. The evoked potential is called transcranial magnetic stimulation-evoked potential.

CONTACTS AND LOCATIONS:
Locations (1):
- Jack Jiaqi Zhang, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided